CLINICAL TRIAL: NCT04939402
Title: SARS-COV-2 Seroprevalence and Seroconversion Among Employees of the Universitair Ziekenhuis Brussel Following COVID-19 Vaccination Using an Adenoviral Vector
Brief Title: SARS-COV-2 Seroprevalence and Seroconversion Among Employees of the UZ Brussel Following COVID-19 Vaccination Using an Adenoviral Vector
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVEMUZ-3
Record Dates: First submitted 2021-04-22; First posted 2021-06-25 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: SARS-CoV-2; Covid19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- General (Other): All patients follow this arm. Patients will undergo 3 blood sample testings at 3 different time points and have to fill in a questionnaire at 3 different time points
  Interventions: Diagnostic Test: Serological testing

INTERVENTIONS:
Diagnostic Test: Serological testing — Antibody testing for Sars-CoV-2 specific antibodies in blood + T cell immunity

SUMMARY:
A novel zoonotic coronavirus was discovered in Wuhan (Hubei Province, China) mid-December 2019 and was named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The virus rapidly spread to the rest of the world, including Europe and explicitly affects the respiratory system, generating Coronavirus disease 2019 (COVID-19).

Employees of the university hospital of Brussels (UZ Brussel) presenting symptoms suggestive of COVID-19 are offered to be tested with real-time PCR on nasopharyngeal swabs. As asymptomatic infections have been described and as the PCR can be negative when taken late after onset of symptoms, serologic tests can be performed. The SARS-CoV 2003 epidemic demonstrated that serological assays were a useful diagnostic tool of non-acute infections. Although it is still uncertain whether convalescing patients have a risk of re-infection, recent data suggest that SARS-CoV-2 antibodies could protect at least for some time from subsequent viral exposures.

As the COVID-19 pandemic had devastating medical, economic and social consequences, safe and effective prophylactic vaccines were urgently needed. And thus several candidate vaccines against SARS-CoV-2 have been developed. The vaccination campaign of the health care workers of the UZ Brussel started mid January 2021. The first available vaccine was the BNT162b2 (Pfizer) vaccine. Early March 2021, in order to accelerate the vaccination of the UZ Brussel employees, the ChAdOx1 nCoV-19 (AZD12222) (Oxford, AstaZeneca) vaccination program was implemented in parallel with the BNT162b2 vaccination program In the COVEMUZ-2 study the investigators have already started to document the SARS-CoV-2 seroprevalence and seroconversion among vaccinated employees (using BNT162b2) in the UZ Brussels.

In this study, the investigators aim to prospectively document the SARS-CoV-2 seroprevalence and seroconversion among vaccinated employees (using ChAdOx1 nCoV-19) of the UZ Brussel, at three different time points, namely 6 weeks (+/- 2 weeks; T1), 6 months (+/- 1 month; T2) and 12 months (+/- 1 month; T3) after the second vaccination.

DETAILED DESCRIPTION:
A novel zoonotic coronavirus was discovered in Wuhan (Hubei Province, China) mid-December 2019 and was named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The virus rapidly spread to the rest of the world, including Europe and explicitly affects the respiratory system, generating Coronavirus disease 2019 (COVID-19).

Employees of the university hospital of Brussels (UZ Brussel) presenting symptoms suggestive of COVID-19 are offered to be tested with real-time PCR on nasopharyngeal swabs. As asymptomatic infections have been described and as the PCR can be negative when taken late after onset of symptoms, serologic tests can be performed. The SARS-CoV 2003 epidemic demonstrated that serological assays were a useful diagnostic tool of non-acute infections. Although it is still uncertain whether convalescing patients have a risk of re-infection, recent data suggest that SARS-CoV-2 antibodies could protect at least for some time from subsequent viral exposures.

As the COVID-19 pandemic had devastating medical, economic and social consequences, safe and effective prophylactic vaccines were urgently needed. And thus several candidate vaccines against SARS-CoV-2 have been developed. The vaccination campaign of the health care workers of the UZ Brussel started mid January 2021. The first available vaccine was the BNT162b2 (Pfizer) vaccine. Early March 2021, in order to accelerate the vaccination of the UZ Brussel employees, the ChAdOx1 nCoV-19 (AZD12222) (Oxford, AstaZeneca) vaccination program was implemented in parallel with the BNT162b2 vaccination program In the COVEMUZ-2 study the investigators have already started to document the SARS-CoV-2 seroprevalence and seroconversion among vaccinated employees (using BNT162b2) in the UZ Brussels.

In this study, the investigators aim to prospectively document the SARS-CoV-2 seroprevalence and seroconversion among vaccinated employees (using ChAdOx1 nCoV-19) of the UZ Brussel, at three different time points, namely 6 weeks (+/- 2 weeks; T1), 6 months (+/- 1 month; T2) and 12 months (+/- 1 month; T3) after the second vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Any adult employee of the UZ Brussel at T1 who has been vaccinated at the UZ Brussel with ChAdOx1 nCoV-19 vaccine between the 2nd of March and the 9th of March 2021 after participating to phase 4 of the COVEMUZ study between the 25th of January and the 12th of February and has provided a signed informed consent.

Exclusion Criteria:

* UZ Brussel employees not active during the inclusion period (T1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To document SARS-CoV-2 seroprevalence among employees of the UZ Brussel after ChAdOx1 nCoV-19 vaccination for SARS-CoV-2, at 8 (+/- 2) weeks after the first vaccination (T1); and 6 and 12 months after the first vaccination (T2 and T3) using a validated immuno-assay for detection of SARS-CoV-2 IgG antibodies
Seroconversion | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To document SARS-CoV-2 seroconversion among employees of the UZ Brussel after ChAdOx1 nCoV-19 vaccination for SARS-CoV-2, at 8 (+/- 2) weeks after the first vaccination (T1); and 6 and 12 months after the first vaccination (T2 and T3) using a validated immuno-assay for detection of SARS-CoV-2 IgG antibodies

SECONDARY OUTCOMES:
SARS-CoV-2 seroprevalence before and after vaccination | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To compare the SARS-CoV-2 seroprevalence before vaccination with the SARS-CoV-2 prevalence after vaccination among employees of the UZ Brussel.
incidence of new definite cases | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To document the incidence of new definite cases of COVID-19 (based on self-reported positive PCR testing on nasopharyngeal swab) among vaccinated employees of the UZ Brussel over a period of a year.
incidence of new probable cases | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To document the incidence of new probable cases of COVID-19 (based on the study questionnaire filled in by the participants) among vaccinated employees of the UZ Brussel over a period of a year.
antibody kinetics of the SARS-CoV-2 specific antibodies using immunassays | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To document the SARS-CoV-2 antibody kinetics after vaccination.
antigen-specificity of the SARS-CoV-2-specific T cells | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To determine the antigen-specificity of the SARS-CoV-2-specific T cells as well as their phenotype and functionality
antibody neutralisation capacity of the SARS-CoV-2 specific B cells using immunassays | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To document the SARS-CoV-2 antibody neutralisation capacity after vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No